CLINICAL TRIAL: NCT01259024
Title: Hepatic Arterial Embolization of Hepatocellular Carcinoma With a Doxorubicin Eluting Bead
Brief Title: The LC Bead Trial; Transarterial Chemoembolization of Hepatocellular Carcinoma (HCC)With a Drug-eluting Bead
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to obtain CMS approval
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201108256
Record Dates: First submitted 2010-11-03; First posted 2010-12-13 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; chemoembolization; transarterial chemoembolization; liver cancer; doxorubicin; drug-eluting beads; LC Bead
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- doxorubicin-eluting LC Bead (Experimental): transarterial chemoembolization using doxorubicin-eluting LC Beads
  Interventions: Device: transarterial chemoembolization using a drug-eluting bead

INTERVENTIONS:
Device: transarterial chemoembolization using a drug-eluting bead — Up to 2 vials of LC Beads will be administered. One 2 mL vial each of 300-500 and 500-700 um LC Beads with 37.5 mg/mL doxorubicin will be prepared and mixed with radiographic contrast. Under fluoroscopic control, the vial of 300-500 um vial will be infused, followed by the vial of 500-700 um LC Beads. If the artery does not reach stasis prior to administration of both vials, and there is residual antegrade flow in the feeding artery, it will be treated with bland embolization similar to chemoembolization.
  Other Names: TACE; DEB TACE

SUMMARY:
This study involves the combined use of the FDA approved device, LC Bead and the FDA approved drug, Doxorubicin for the treatment of primary hepatocellular carcinoma (HCC). The current indication of the LC Bead is for the embolization of hypervascular tumors and arteriovenous malformations. The study is designed to establish if drug eluting beads are more effective and less toxic than standard chemoembolization treatment.

DETAILED DESCRIPTION:
Patients will be given IV fluids and premedication with 500 mg metronidazole, 10 mg dexamethasone, and 8 mg ondansetron to prevent infection, limit pain and nausea. The femoral artery will be accessed and a catheter advanced into the superior mesenteric artery. Positioning of all catheters will be confirmed by injection of radiographic contrast material. Superior mesenteric angiography will be performed with images obtained through the portal venous phase to confirm patency and flow direction of the portal vein and determine the presence of aberrant supply to the right lobe of the liver by the superior mesenteric artery. The catheter will then be advanced into the celiac artery. Celiac angiography will be performed to determine remainder of the hepatic arterial anatomy. Selection of the tumor bearing artery will then be performed with a microcatheter which is advanced through the catheter in the celiac artery origin. Selection will be guided by fluoroscopy and will be at the lobar level or peripherally in all cases. Once the feeding vessel has been selected and confirmed by contrast injection, the physician will initiate embolization with LC Beads. Up to two vials of LC Beads will be administered. One 2 mL vial each of 300-500 and 500-700 um LC Beads with 37.5 mg/mL doxorubicin will be prepared. The LC Beads will be mixed with radiographic contrast to ensure fluoroscopic visibility during injection. Under careful fluoroscopic control, the vial of 300-500 um vial will be infused, followed by the vial of 500-700 um LC Beads. If the artery reaches stasis prior to administration of both vials, the residual volume of LC Beads will be noted on the surgical report form. If after administration of the DEB, there is residual antegrade flow in the feeding artery, it will be treated with bland embolization similar to chemoembolization. After confirming that the artery is appropriately treated, all catheters and guidewires will be removed from the femoral artery and hemostasis obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patent main portal vein with hepatopetal flow
* Bilirubin less than or equal to 2.5 mg/dl, albumin >2.8g/dl, alkaline phosphatase <630IU/L, AST <235IU/L, ALT <265IU/L, INR <2.0, PTT <40sec., absolute neutrophil count >1K/cumm, platelet count >100K/cumm
* No encephalopathy
* No previous biliary ductal intervention
* Child A status
* Confirmation of Hepatocellular Carcinoma (through biopsy or radiological exam)
* Unresectable HCC and ineligible for possible curative therapies
* Normal ECG with QT <480 msec within the previous 2 months
* Normal MUGA scan within the previous 2 months
* Measureable disease per the Response Evaluation Criteria in Solid Tumors (RECIST)
* Subject is competent and willing to provide written informed consent in order to participate in the study

Exclusion Criteria:

* Thrombosis or hepatofugal flow in the main portal vein; presence of a large shunt which in the operator's opinion precludes embolization
* Replacement of greater than 50% of the liver parenchyma by tumor
* Bilirubin greater than or equal to 2.6 mg/dl
* ECOG performance status of 2 or greater
* Previous liver directed therapy
* Previous biliary intervention (excluding cholecystectomy)
* Allergy to iodinated contrast used for angiography
* Elevated creatinine greater than or equal to 1.8 mg/dl
* Women who are pregnant or nursing
* Patients in which any of the following are contraindicated: 1)the use of doxorubicin, 2)MRI or CT scans, 3) Hepatic embolization procedures
* Patients with active bacterial or fungal infection that is deemed to be clinically significant by the investigator
* Patients with cardiac disease, including congestive heart failure, recent myocardial infarction, or uncontrolled arrhythmias
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nael E. Saad, M.D., Principal Investigator — Mallinckrodt Institute of Radiology/Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital/Washington Univesity School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dhanasekaran R, Kooby DA, Staley CA, Kauh JS, Khanna V, Kim HS. Comparison of conventional transarterial chemoembolization (TACE) and chemoembolization with doxorubicin drug eluting beads (DEB) for unresectable hepatocelluar carcinoma (HCC). J Surg Oncol. 2010 May 1;101(6):476-80. doi: 10.1002/jso.21522. PMID 20213741
- [Background] Biselli M, Andreone P, Gramenzi A, Trevisani F, Cursaro C, Rossi C, Ricca Rosellini S, Camma C, Lorenzini S, Stefanini GF, Gasbarrini G, Bernardi M. Transcatheter arterial chemoembolization therapy for patients with hepatocellular carcinoma: a case-controlled study. Clin Gastroenterol Hepatol. 2005 Sep;3(9):918-25. doi: 10.1016/s1542-3565(05)00425-8. PMID 16234031
- [Background] Malagari K, Pomoni M, Kelekis A, Pomoni A, Dourakis S, Spyridopoulos T, Moschouris H, Emmanouil E, Rizos S, Kelekis D. Prospective randomized comparison of chemoembolization with doxorubicin-eluting beads and bland embolization with BeadBlock for hepatocellular carcinoma. Cardiovasc Intervent Radiol. 2010 Jun;33(3):541-51. doi: 10.1007/s00270-009-9750-0. Epub 2009 Nov 24. PMID 19937027
- [Background] Namur J, Wassef M, Millot JM, Lewis AL, Manfait M, Laurent A. Drug-eluting beads for liver embolization: concentration of doxorubicin in tissue and in beads in a pig model. J Vasc Interv Radiol. 2010 Feb;21(2):259-67. doi: 10.1016/j.jvir.2009.10.026. PMID 20123210
- See also: Interventional Radiological Treatment of Hepatocellular Carcinoma — http://www.medscape.com
- See also: Drug-Eluting Beads Significantly Reduce Doxorubicin Toxicity in Patients With HCC — http://www.docguide.com
- See also: Efficacy of Drug-Eluting Beads in Chemoembolization of Hepatocellular Carcinoma — http://www.projectsinknowledge.com
- See also: Chemoembolization using Drug Eluting Beads is an effective procedure with a favourable pharmacokinetic profile — http://www.biocompatibles.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant was screened and recruited on 1/5/2012
Pre-assignment Details: Single-arm study - participant received 1st trans-arterial chemoembolization treatment on 1/23/2012, second treatment on 2/20/2012, and third treatment on 3/20/12. Physician decision to withdraw participant on 4/12/2012 due to denial of CMS reimbursement.
Period: Overall Study
Arm/Group | Doxorubicin-eluting LC Bead
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Doxorubicin-eluting LC Bead
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: To Collect Data on Patients With Hepatocellular Carcinoma (HCC) Being Treated With Chemoembolization With Doxorubicin Eluting Beads (DEB).
Description: 4-6 weeks after initial treatment, follow-up imaging will be obtained. With positive response to treatment, follow-up imaging will be obtained every 12 weeks. If a new tumor develops or if local progression of the treated malignancy occurs, the patient may be retreated with LC Beads 4-6 weeks after the first treatment with re-imaging 4-6 weeks following each subsequent treatment.
Time Frame: Patients will participate in protocol until date of death, liver transplantation, or withdrawal from study.
Population: One participant was enrolled on this IDE and was treated on protocol for 14 weeks. After being made aware that CMS would not provide reimbursement, the PI decided to withdraw the patient and continued to treat off protocol.
Arm/Group | Doxorubicin-eluting LC Bead
Number analyzed (Participants) | 0

2. Primary Outcome: Determine Efficacy (Based on Whether the Study is Positive or Negative) of the Embolization With the LC Bead in Treatment of HCC With Imaging Outcomes Using Modified RECIST and EASL Criteria.
Description: as for outcome 1
Time Frame: Patients will participate in protocol until date of death, liver transplantation, or withdrawal from study.
Population: 1 patient was enrolled in the study, but was withdrawn by the PI due to inability to obtain CMS reimbursement. The patient was treated off protocol and therefore there are no study results to be analyzed.
Arm/Group | Doxorubicin-eluting LC Bead
Number analyzed (Participants) | 0

3. Primary Outcome: Monitor Safety After Treatment of DEB by Measuring Liver Function Tests and Assessing Performance Status.
Description: as for outcome 1
Time Frame: Patients will participate in protocol until date of death, liver transplantation, or withdrawal from study.
Arm/Group | Doxorubicin-eluting LC Bead
Number analyzed (Participants) | 0

4. Secondary Outcome: To Track Survival Following Treatment With DEB to Confirm That Any Gains in Response Are Associated With an Increase in Survival.
Description: as for outcome 1
Time Frame: Patients will participate in protocol until date of death, liver transplantation, or withdrawal from study.
Population: 1 participant was enrolled, analyzed was 0.
Arm/Group | Doxorubicin-eluting LC Bead
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 14 weeks, then participant was withdrawn
Arm/Group | Doxorubicin-eluting LC Bead
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin-eluting LC Bead (N=1)
fatigue (General disorders) | 1 (1) — generalized fatigue
right groin burning pain (Injury, poisoning and procedural complications) | 1 (1) — Burning to right groin with post-procedure hematoma
back pain (General disorders) | 1 (2) — low back pain
anorexia (Gastrointestinal disorders) | 1 (2) — anorexia
nausea (Gastrointestinal disorders) | 1 (1) — nausea

LIMITATIONS AND CAVEATS:
Overall limitation was related to not reaching the target number of participants needed to achieve target power and statistically reliable results due to denial of CMS reimbursement. Majority of this patient population is covered by CMS services.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes